CLINICAL TRIAL: NCT05169281
Title: Cluster Randomized Trial of a Mailed At-home Kit on Disposal of Unused Opioids Following Surgery
Brief Title: Distribution of Medication Disposal Packets - Acute Opioid Prescribing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Anish Agarwal, MD, MPH, MS, Assistant Professor & Chief Wellness Officer | Department of Emergency Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 827461_1
Record Dates: First submitted 2021-11-19; First posted 2021-12-23 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Orthopedic Surgery; Neurosurgery; Surgery; Opioid Use; Opioid Misuse
Keywords: Opioid Prescribing; Mobile Health; Quality Improvement; Learning Health Systems
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant will be blinded to their random assignment into the control or treatment (medication disposal packet) group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual care consisted of a text message hyperlink to nearby disposal locations.
- Intervention (Experimental): Intervention participants were mailed an at-home disposal packet timed to arrive between post-operative days four and seven based on prior data collection on reported use.
  Interventions: Other: Medication Disposal Packet

INTERVENTIONS:
Other: Medication Disposal Packet — The disposal packet (DisposeRx Inc.) contains a powder that sequesters unused opioids in a polymer gel. The kits reached patients four days following their surgery based on prior data to leverage availability bias, or a tendency to think or act on things that are most present in one's mind, and provided patients with a disposal technique when they were likely to be finished with their opioids. The process of mailing the disposal packet is simple, low cost (~$1.50/ mailed packet) and scalable.
  Arms: Intervention

SUMMARY:
Many prescription opioids following surgery are left unused and are at risk of being misused or diverted. Encouraging proper disposal is important, yet motivating this behavior remains challenging as patients must understand the risks of opioids, the benefits of disposal, and identify opportunities and places to dispose of them safely. Alternative disposal techniques can improve disposal rates but may be lost or forgotten. Applying behavioral economics techniques may lower the barriers and promote disposal. The objective is to test the effect of a specifically timed, mailed, at-home kit on disposal rates following surgery.

DETAILED DESCRIPTION:
A pragmatic, cluster-randomized quality improvement study embedded in an existing automated, post-operative text messaging program to capture patient-reported outcomes (e.g., pain score, opioid use, ability to manage pain) and disposal as part of usual care. It was approved by the University of Pennsylvania Institutional Review Board with a waiver of informed consent.

All patients, 18 years or older, undergoing an orthopedic or urologic procedure and prescribed an opioid were approached and consented via text messaging. Patients without access to a text message capable device or non-English speaking were excluded. Participants were block randomized to usual care or a mailed at-home disposal packet. Usual care consisted of a text message hyperlink to nearby disposal locations. Intervention participants were mailed an at-home disposal packet timed to arrive between post-operative days four and seven based on prior data collection on reported use. The disposal packet (DisposeRx Inc.) contains a powder that sequesters unused opioids in a polymer gel. Patients self-reported disposal via the automated system.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 or older
* Undergoing an orthopedic or urologic procedure
* Prescribed an opioid
* SMS capable mobile device
* English speaking

Exclusion Criteria:

* Under 18
* Does not own a text message capable mobile phone
* non-English speaking

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 657 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Self-Reported Opioid Disposal | The duration of the study; two months
  The opioid disposal kits provided patients with a timely, easy, and safe disposal technique which was sent to them between post-operative day 4-7 which corresponds with historical trends in declining opioid use. This primary outcome is self-reported opioid disposal which is obtained via an automated text message sent to patients on post operative day 7.

CONTACTS AND LOCATIONS:
Overall Officials: Anish Agarwal, MD, Principal Investigator — University of Pennsylvania; Daniel Lee, MD, Principal Investigator — University of Pennsylvania; Zarina Ali, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be shared.

REFERENCES:
- [Background] Hill MV, McMahon ML, Stucke RS, Barth RJ Jr. Wide Variation and Excessive Dosage of Opioid Prescriptions for Common General Surgical Procedures. Ann Surg. 2017 Apr;265(4):709-714. doi: 10.1097/SLA.0000000000001993. PMID 27631771
- [Background] Bicket MC, Long JJ, Pronovost PJ, Alexander GC, Wu CL. Prescription Opioid Analgesics Commonly Unused After Surgery: A Systematic Review. JAMA Surg. 2017 Nov 1;152(11):1066-1071. doi: 10.1001/jamasurg.2017.0831. PMID 28768328
- [Background] Kennedy-Hendricks A, Gielen A, McDonald E, McGinty EE, Shields W, Barry CL. Medication Sharing, Storage, and Disposal Practices for Opioid Medications Among US Adults. JAMA Intern Med. 2016 Jul 1;176(7):1027-9. doi: 10.1001/jamainternmed.2016.2543. No abstract available. PMID 27295629
- [Background] Brummett CM, Steiger R, Englesbe M, Khalsa C, DeBlanc JJ, Denton LR, Waljee J. Effect of an Activated Charcoal Bag on Disposal of Unused Opioids After an Outpatient Surgical Procedure: A Randomized Clinical Trial. JAMA Surg. 2019 Jun 1;154(6):558-561. doi: 10.1001/jamasurg.2019.0155. PMID 30916733
- [Background] Agarwal Anish K., Ali Zarina S., Sennett Brian, et al. An Automated Text Messaging Program to Inform Postoperative Opioid Prescribing. NEJM Catal [Internet] [cited 2021 Feb 18];2(3). Available from: https://doi.org/10.1056/CAT.20.0440
- [Background] Agarwal AK, Lee D, Ali Z, Sennett B, Xiong R, Hemmons J, Spencer E, Abdel-Rahman D, Kleinman R, Lacko H, Horan A, Dooley M, Hume E, Mehta S, Delgado MK. Patient-Reported Opioid Consumption and Pain Intensity After Common Orthopedic and Urologic Surgical Procedures With Use of an Automated Text Messaging System. JAMA Netw Open. 2021 Mar 1;4(3):e213243. doi: 10.1001/jamanetworkopen.2021.3243. PMID 33764425